CLINICAL TRIAL: NCT07365761
Title: Emotional Assessment and Tiered Individualized Psychological Support for Newly Diagnosed Postoperative Gynecologic Patients: Development and Testing of the E-MOTE Artificial Intelligence Robot
Brief Title: Emotional Assessment and Tiered Individualized Psychological Support of the Artificial Intelligence Robot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202504008RINC
Record Dates: First submitted 2025-07-25; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Emotional Assessment; Nursing; Gynecological Cancers
Keywords: Artifical inteligence; Robot; Emotional assessment; Psychological support; Nursing

STUDY DESIGN:
Intervention Model Description: This intervention module will first classify different levels of emotional distress using the Distress Thermometer, then provide corresponding dialogue modules tailored to the severity. These will be accompanied by emotion-generated empathetic conversations for deeper engagement, followed by a guided session of self-affirmation relaxation training. Subsequently, a Q&A session on the self-affirmation relaxation training will be conducted to reinforce the practice.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine care
- Intervention Group (Experimental): The intervention group will receive the E-MOTE robot, which conducts emotional assessments, and provides a session of self-affirmation relaxation training followed by a Q&A session.
  Interventions: Other: E-MOTE group

INTERVENTIONS:
Other: E-MOTE group — Participants in the experimental group will receive the E-MOTE robot intervention on the first and second days after surgery. The intervention includes an emotional assessment, followed by appropriate dialogue modules tailored to the level of emotional distress. These are supplemented with emotion-generated empathetic conversations for deeper engagement, a session of self-affirmation relaxation training, and a subsequent Q&A session.
  Arms: Intervention Group

SUMMARY:
To develop the E-MOTE robot and evaluate its effectiveness in addressing psychological distress, physical symptom, stress index, and quality of life, as well as to explore its clinical applicability.

DETAILED DESCRIPTION:
This study is grounded in the Social Cognitive Theory of Self-Regulation as its theoretical framework and aims to develop a robot equipped with functions of Emotion, Monitor, Optimize, Tailor, and Engage (E-MOTE). The intervention is designed to support newly diagnosed gynecological cancer patients in more effectively managing their emotions throughout the surgical treatment process, with the goal of positively influencing symptom management and quality of life.At the same time, the investigators will conduct qualitative interviews with nursing staff to understand their perceptions and thoughts about the robot.

ELIGIBILITY:
Stage 1 (For patients and nurse) ***Patients***

Inclusion Criteria:

* Aged 18 years or older.
* Diagnosed with gynecologic cancer and undergoing surgery.
* Willing to receive E-MOTE robot and wear a smart wearable device.
* Willing to complete pre-test and post-test questionnaires.

Exclusion Criteria:

* Unable to communicate clearly.
* Unwilling or unable to participate in the study in its entirety.

***Nurse***

Inclusion Criteria:

* Aged 18 years or older.
* As a clinical nurse and has cared for patients who received the E-MOTE robot

Exclusion Criteria:

- Unwilling to participate in the qualitative interview.

Stage 2 (only for patients) ***Intervention group***

Inclusion Criteria:

* Aged 18 years or older.
* Diagnosed with gynecologic cancer and scheduled to undergo surgery.
* Willing to receiveE-MOTE robot and to wear a smart wearable device.
* Willing to complete pre-test and post-test questionnaires.

Exclusion Criteria:

* Unable to communicate clearly.
* Unwilling or unable to participate in the study in its entirety.

***Control group***

Inclusion Criteria:

* Aged 18 years or older.
* Diagnosed with gynecologic cancer and scheduled to undergo surgery.
* Willing to complete pre-test and post-test questionnaires.

Exclusion Criteria:

* Unable to communicate clearly.
* Unwilling or unable to participate in the study in its entirety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Distress | Measurements will be taken before the intervention, three days after surgery, and one week after discharge.
  Investigators utilized the Distress Thermometer(DT) as the primary outcome measure. The scale uses a 11 Liker scale, where 0 indicates no distress at all and 10 represents the most severe distress.Higher score indicates a more severe distress. When the score is 4 or higher, a Problem List (PL) is used to further identify factors contributing to the emotional distress.
Depression | Measurements will be taken before the intervention, three days after surgery, and one week after discharge.
  Investigators utilized the Patient Health Questionnaire (PHQ-9) as the primary outcome measure to assess depression. The scale consists of 9 items, each rated on a 4-point Likert scale (0 = not at all, 3 = nearly every day). The total score ranges from 0 to 27, and depression severity can be categorized as mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20 or above).Higher score indicates a more severe depression.

SECONDARY OUTCOMES:
Usability of the robot | Measurements will be taken three days post-surgery.
  Investigators used Bot Usability Scale(BUS) to asses the usability of the robot. The scale consists of 15 items, each rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree), higher score indicates greater usability.
Quality of Life Measurement | Measurements will be taken before the intervention, three days after surgery, and one week after discharge.
  Investigator use the partial itmes of European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30) to measure quality of life. These two item is scored on a scale from 1 to 7, with higher scores indicating better quality of life.
Loneliness | Measurements will be taken before the intervention, three days after surgery, and one week after discharge.
  Investigators utilized the Caring Loneliness Scale to assess loneliness. The scale consists of 24 items, each rated on a 5-point Likert scale (1 = never, 5 = always), with higher scores indicating greater feelings of loneliness.
Symptom Severity | Measurements will be taken before the intervention, three days after surgery, and one week after discharge.
  Investigators utilized the Numerical Rating Scale to assess participants' subjective experiences by measuring the severity of various symptoms over the past week. Each symptom was rated on a scale from 0 to 10 (0 = no symptoms at all, 10 = the worst severity the participant can imagine). Higher score indicate more severity. This items included difficulty urinating, lower limb lymphedema, hot flashes caused by premature menopause, and perineal dryness.
Physiological objective indicators | Measurements will be taken before the intervention, three days after surgery, and one week after discharge.
  Objective physiological indicators were measured using wearable smart wristbands, including heart rate, heart rate variability, and stress index.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided